CLINICAL TRIAL: NCT06420544
Title: Japi: Cognitive, Emotional and Social Stimulation for Preschool Children
Acronym: Japi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: University of Talca (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Principal Investigator, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FONDEF ID22I10126
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Behavioral Problem of Child
Keywords: Executive Functions; Behavioral Problem; Children; Videogame; Non-cognitive skills; Cognitive skills
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Acceptability, feasibility and efficacy of this intervention will be measured, including the measurement of outcomes (skill formation) compared with a 'placebo' control group among pre-school children from low socio-economic backgrounds in Santiago. A mixed-method design with a strong qualitative component to understand better the factors that might facilitate or interfere with the delivery and acceptability of this intervention will be conducted. At the start of the study there will be a mapping the structure of the schools, the locations, staff composition, characteristics of the children and families, and other contextual factors important for the successful implementation of the intervention.
  Schools that fulfil the inclusion and exclusion criteria will be invited to participated. Six schools be selected and will be randomized and allocated in 1:1 proportion to intervention and control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The whole intervention has 24 sessions. Children will play with the game two times a week, each lasting 15 minutes, over a period of 12 weeks. Each session stimulates two skills (one cognitive and one non-cognitive skills) and has eight activities with increasing levels of difficulty.
  Interventions: Behavioral: JAPI: Cognitive, Emotional and Social Stimulation for Preschool Children
- Control group (No Intervention): The control group receives standard school curricula, which is not a manualized intervention. The standard curriculum is provided by the Ministry of Education with a guideline called "Curricular Bases for Kindergarten Education" which includes pre-kindergarten directions to Early Year Educators regarding emotion regulation and planification to implement in class.

INTERVENTIONS:
Behavioral: JAPI: Cognitive, Emotional and Social Stimulation for Preschool Children — Those children in the intervention group will play with the gaming platform "Japi" using a tablet device in a designated time given from schools' authorities. Early Year Educators will be present to help with the discipline and motivation of the students and Research Assistants will be there as well to provide technical support for the use of the equipment.
  The intervention has 24 sessions, and the dosage will be two sessions of 15 minutes each per week for 12 weeks. Sessions number 1 to number 8 are focused on emotional regulation and inhibitory control. Sessions number 9 to 16 work on working memory and problem-solving. Sessions number 17 to 24 promote empathy and planification skills. Each session will have eight activities with increasing levels of difficulty.
  Other Names: JAPI
  Arms: Intervention group

SUMMARY:
Mental health disorders are one of the leading causes of illness globally, and their relevance is expected to increase. Low and Middle Income Countries (LMIC), already facing psychological and behavioral issues due to chronic adversity, were further impacted during the COVID-19 pandemic. A study showed that symptoms of depression and anxiety in youth doubled during the first year of the pandemic compared to the pre-pandemic period.

A study in China found that the prevalence of the total difficulties was (8.2%), with conduct problems (7.0%), peer problems (6.6%), and hyperactivity-inattention (6.3%) among the most prevalent. In this study emotional problems reached 4.7%. Finally, recent evidence has revealed that students' psychosocial and behavioral problems have increased in the early stage of schools reopened. Several international agencies have calls on governments, and public and private sector partners, to commit, communicate and act to promote mental health for all children, protect those in need of help, and care for the most vulnerable.

The importance of psychosocial skills acquired in early childhood, such as emotional regulation and social problem-solving, for preventing mental disorders was highlighted. Studies indicate that the development of executive functions and non-cognitive skills in early childhood has a positive impact on long-term health and economic productivity.

However, the treatment gap for mental disorders in LMIC is significant, with only one in ten affected receiving treatment. Preventive interventions are needed, particularly in early childhood, to improve cognitive and socio-emotional skills.

Objective: The research proposal aims to develop a gaming platform aiming to improve cognitive and non-cognitive skills in early childhood at schools with high socio-economic vulnerability, supported by Early Years Educators and Parents using a dashboard integrated in a whole system housed in local server, and to evaluate the acceptability and feasibility of this gaming platform and dashboards, with the ultimate goal of reducing behavioral problems, and improving functional and performance outcomes later in life.

Outcomes: Acceptability; Feasibility; Cognitive and non-cognitive skills; Working Memory; Inhibitory control; Emotion recognition; Social competence; Behavioral problems and psychological assessment.

DETAILED DESCRIPTION:
Problem and opportunity:

Mental health disorders are among the leading causes of the Global Burden of Disease, and their relative importance is predicted to rise globally. Adversity is one of the most important risk factors associated with an increased incidence of psychological and behavioral problems. Acute or chronic adversity is common in Low and Middle Income Countries (LMIC) settings and unsurprisingly, psychological and behavioral problems are highly prevalent in LMIC, which have to deal with these emerging problems with scarce resources. During the COVID-19 pandemic, this scenario has worsened globally. One recent systematic review has showed that pooled estimates obtained in the first year of the COVID-19 pandemic suggest that 25.2% (95% Confidence Interval (CI), 21.2%-29.7%) of youth globally are experiencing clinically elevated depression symptoms, while 20.5% (95% CI, 17.2%-24.4%) of youth are experiencing clinically elevated anxiety symptoms. These pooled estimates, which increased over time, are double of pre pandemic estimates. And regarding behavioral problems, a study in China found that the prevalence of the total difficulties was (8.2%), with conduct problems (7.0%), peer problems (6.6%), and hyperactivity-inattention (6.3%) among the most prevalent. In this study emotional problems reached 4.7%. Finally, recent evidence has revealed that students' psychosocial and behavioral problems have increased in the early stage of schools reopened. Several international agencies have calls on governments, and public and private sector partners, to commit, communicate and act to promote mental health for all children, protect those in need of help, and care for the most vulnerable. The State of the World's Children 2021, UNICEF's most comprehensive look at the mental health of children in the 21st century, calls on "urgent investment in child and adolescent mental health across sectors, not just in health, to support a whole-of-society approach to prevention, promotion and care" and "integrating and scaling up evidence-based interventions across health, education and social protection sectors […]; and ensuring schools support mental health through quality services and positive relationships".

Along with the magnitude of the problem, the treatment gap for mental health disorders is large: one in every ten people with mental disorders receives treatment in LMIC. The ideal strategy to tackle this gap should be that of preventing the onset of these conditions. Most adult mental disorders start in childhood or adolescence, and delaying or preventing the onset can have a substantial impact. However, few preventive interventions or interventions to increase resilience to adversity have been developed, and even fewer tested in LMIC. There is evidence to suggest that strengthening cognitive and socio-emotional skills might result in a reduced incidence of mental disorders. For instance, reduced emotional regulation, and poor social problem-solving have been associated with increased incidence of depression.

Basic psychological skills acquired early in life have been associated with a range of important social and economic outcomes later in life. Early childhood is a critical time for psychosocial development. Until recently, years of education and Intelligence Quotient (IQ) were the main measures to assess the relationship between human capital and economic development. More recently, researchers have acknowledged that skills such as maintaining good interpersonal relations, controlling impulses, or demonstrating goal-directed behavior are critical to physical and mental health and economic productivity. The Nobel prize economist, James Heckman, highlighted the importance of these skills, which he originally called non-cognitive skills, for economic development. Scientific evidence has recently indicated that the stimulation of cognitive and non-cognitive skills in the first years of life promotes general development and has a beneficial long-term impact on health and on different economic indicators . However, much of this evidence comes from studies in the United States, Europe of other develop countries, such as the High/Scope Perry Preschool Study, the Abecedarian Project , Head Start, and Early Head Start. Many of these interventions were costly and difficult to implement.

Several studies have investigated how the capacity to regulate emotions and behaviors is associated with social, health, educational, and labor outcomes. Studies from neurobiology to behavioral economics show that emotions affect a person's ability to self-regulate and that this, in turn, affects cognitive skills and subsequent self-regulatory capacity. Executive functions, involving the regulation and control of cognitive processes, are closely linked to skills leading to better problem solving, task persistence, self-esteem, school performance, and better social adjustment with a reduction in aggressive and other behavioral problems. Healthy development of executive functions early in life predicts better self-regulatory capacity later. The growing scientific knowledge-based emotional self-regulation or social skills linked to the developing brain can be leveraged to engender new intervention approaches. There is significant evidence that structural and functional plasticity in many brain core centers involved in executive functions and self-regulatory processes develops rapidly during early childhood. Most of the evidence to support the association between early acquired psychosocial skills and functional outcomes later in life comes from developed countries. There is a need to replicate these findings in resource-poor settings.

In addition, the evidence suggests that children from low-income families may begin the preschool stage with less development of academic (such as pre-calculus and initial language) and non-academic skills (such as emotional, social, and health competence in general) when compared with children from higher-income families. These differences would contribute to the increase in socio-emotional, educational, and health disparities in the long term. Add to this the evidence that critical aspects of human development occur between 3 and 7 years, such as the recognition of emotions, the control of behavior, and the development of Executive Functions, it is essential to work with children who have greater economic vulnerability and to stimulate these skills early.

As our approaches become more interdisciplinary, several important questions arise: What is the effect of improving psychosocial skills on health, educational, and economic outcomes? What interventions are most effective at bolstering these functions and abilities? What is the applicability of such interventions across diverse cultural groups and in low-resource settings? Valid and reliable measures to assess these skills are lacking, especially for use in less developed countries. Furthermore, it would be important to incorporate more objective neurocognitive and physiological variables into the study of these regulatory processes. A concerted effort is needed to identify these critical psychosocial skills that can be incorporated into interventions to improve children's wellbeing globally. Multi-disciplinary research efforts can advance our understanding of these essential elements of human capital formation and their role in social and economic success in diverse settings.

The penetration of new technologies (smartphones, tablets, wearable devices) is increasing all over the world and opening unimaginable opportunities to advance this field, especially due to the effect of the covid-19 pandemic. Technological platforms offer an incredible opportunity to reach out to underserved and remotely located populations. The use of smartphones and tablets is increasing at a fast speed in most LMIC. These devices allow us to use more sophisticated software as well as all 'old' functionalities such as text messaging or live telephony. Gaming offers an excellent opportunity to engage young kids and deliver early life interventions at a low cost and at a large scale. The use of games in the educational sector is wide and continues to grow. There is good evidence that the use of technology among pre-school kids is feasible and growing. There are already recommendations of the features that apps need to have to promote learning and creativity. No other tablet games for young children are known that aim to stimulate multiple skills (working memory or inhibitory control, self-regulation, and social problem solving) with a single unified game. Other than teaching skills, technology might also allow capturing large amounts of data, which can help at the same time with one piece of software us understand better the mechanisms whereby skills are learned and the pathways to larger impact later in life. If these interventions effectively strengthen skills vital to improve health, social, and economic outcomes, the gains for society could be substantial. A large number of applications have been launched, though very few tested, to prevent mental disorders or behavioral problems. However, there is a marked paucity in the development of preventive interventions delivered via technology, especially early in life. There are a few games to foster specific psychosocial skills among pre-school children but comprehensive platforms that stimulate diverse functions, such as working memory, inhibitory control, emotion recognition or social competence, are not available.

Latin America has been a leading region pioneering initiatives aiming to stimulate basic psychosocial skills early in life. In Chile, programs to encourage mothers to stimulate the psychosocial skills of their children started in the seventies but the initial interest somehow lost impetus for political and economic reasons. More recently, as part of a major World Bank project in which members of our group participated, parents of low socioeconomic status were trained to improve the skills of their young children (aged <=5). Our group also undertook a large Randomized Controlled Trail (RCT) of a mental health school intervention for adolescents. One of the main lessons of this study was the need to focus on interventions at earlier ages to prevent rather than treat mental health problems. There is also evidence from other Chilean school programs that psychosocial skills are associated with better educational outcomes. Overall, there is consensus that in spite of the importance of the topic, there has been little research from LMICs. This proposal brings together a wide range of expertise across multiple disciplines including psychology, neuroscience, epidemiology, intervention trials, education, and economics. New methods and technologies are also being incorporated into this proposal. Developing effective early life interventions and assessing the mechanisms leading to changes using top-of-the-range, non-invasive technology are key features of this proposal. The results of this research will lay the foundations for future programs to learn how young children acquire skills, how the developing brain works, whether or not these skills predict future outcomes, and how these interventions can be scaled up.

Pandemic effect on tech use:

The digital revolution is evolving with an unprecedented explosion of technology development to transform mental health care delivery, with its emphasis on computing power and mobile technology. These platforms are becoming the medium through which assessment and intervention are taking place. The COVID-19 crisis has fast forwarded the use of technology in mental health care; therefore, it is crucial to scale up access to mental health interventions during and after COVID-19.

Taking all into account, the general objective of this study is to develop a gaming platform aiming to improve cognitive and non-cognitive skills in early childhood at schools with high socio-economic vulnerability, supported by Early Years Educators and Parents using a dashboard integrated in a whole system housed in local server, and to evaluate the acceptability and feasibility of this gaming platform and dashboards, with the ultimate goal of reducing behavioral problems, and improving mental health and functional and performance outcomes later in life.

ELIGIBILITY:
For schools:

Inclusion criteria:

1. Schools located in Santiago (Chile).
2. Schools with Preschool Education.
3. Mixed-sex schools.
4. Schools with vulnerability (≥75%), measured with the School Vulnerability Index - National System of Equality Allocation (IVE-SINAE). This index is the proportion of students in a given school with high vulnerability. This index considers the following socioeconomic variables to group the schools: mother's educational level, father's educational level, and total monthly household income, among others.

Exclusion criteria:

1. Three or more classes in Preschool. This criterion was considered for economic and practical reasons.
2. Implementing a manualized program to promote cognitive or social-emotional skills.
3. Participating in a similar study.

For students:

Inclusion criteria:

1) Children attending pre-kindergarten

Exclusion criteria:

1. Children with intellectual disability
2. Children unable to understand and speak Spanish

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability: Early Year Educators | through study completion, an average of 6 month
  Acceptability will be evaluated using one questionnaire that will be answered every week by the Early Year Educators (EYE). It will include questions regarding the fidelity of the implementation (e.g. "How many sessions children were able to play during the week?" "Be the panel to know the progress of the children?" "How many minutes were used to support each child during the week?", "Was the activity in this session interesting/relevant?" They also ask about the things they liked about the sessions and what they would change; and specifically, for EYE: "was feedback given to parents to promote the use of the gaming platform?"). The team will also solicit feedback on possible changes to be included in the future (e.g. "Is there anything that would be changed/replaced/included?").
Acceptability: Students | through study completion, an average of 6 month
  A brief assisted survey will also be carried out on the students, carried out in the middle and at the end of the intervention to assess if a children liked the intervention.
Feasibility of the intervention: Recruitment | through study completion, an average of 6 month
  Data will be collected on the number of schools that are eligible, those that are contacted, and those that agree to participate. Data will also be collected on the number of students, parents, and Educators contacted and those who consent and agree to participate.
Feasibility of the intervention: Assesment parameters | through study completion, an average of 6 month
  Data will also be collected on the time needed to complete the questionnaires and student assessment tests, and the loss of participants during follow-up.
Feasibility of the intervention: Progress on the videogame | through study completion, an average of 6 month
  Automated data on the use of the game (number of sessions played, activities completed and level reached) will be captured via a server in those 3 schools with intense EYE support.

SECONDARY OUTCOMES:
Working Memory: Corsi Block Test | through study completion, an average of 6 month
  This test assesses visuo-spatial short-term working memory. It involves repeating a sequence of up to nine identical spatially separated blocks on a screen. The sequence starts out simple but becomes more complex until the subject's performance begins to decline. This number is known as the Corsi Span. The higher score the better the skill.
Working Memory: Auditive Working Memory test | through study completion, an average of 6 month
  A sequence of audio messages of increased difficulty is presented, and the child is requested to remember these messages. The higher score the better the skill.
Inhibitory control: The Hearts and Flowers task | through study completion, an average of 6 month
  The Hearts and Flowers task is a hybrid combining elements of Simon and spatial Stroop tasks. For congruent trials, subjects are to obey the rule, "Press on the same side as the stimulus (Hearts)." For incongruent trials, subjects are to follow the rule, "Press on the side opposite the stimulus (Flowers)." It requires working memory and inhibition control. The higher score the better the skill.
Emotion recognition: Assessment of Children's Emotions Skills | through study completion, an average of 6 month
  It consists of facial expressions task aiming to evaluate emotion expression knowledge and whether the subjects exhibit any anger bias. The 26-item scale consists of colour photographs of ethnically diverse elementary schoolchildren depicting four expressions of each of the four basic emotions (happy, sad, angry, and scared) and 10 images of children without obvious facial expressions. The examiner shows the child the photographs one at a time and each time asks, "Is the child in the picture happy, sad, angry, or scared?" Then the examiner registers the child's answer. The emotion accuracy score reflects how many items the children answer correctly, and the anger bias score is the percentage of time the children incorrectly identify the faces as displaying anger. The higher score the better the skill.
Social competence: Challenging Situations Task | through study completion, an average of 6 month
  This instrument evaluates the ability of children to solve social problems. The children are presented six vignettes that describe problems between peers. Following the presentation of each challenging situation, four pictures of happy, sad, angry, and neutral affect are presented in random order. The child is asked to point to the picture that best describes how they feel when [this situation] happens. Then four pictures of behavioral responses (prosocial, aggressive, manipulation of others' feelings, and avoidant) are presented in random order and the child is asked "What do in this situation]?" The answers are categorized into four possibilities: prosocial, aggressive, cry, and avoidant. Scores for affective and behavioral responses used are the number of times each affect and each behavioral response is chosen by each child across the six situations. The higher score the better the skill.
Social competence: The Social Competence Scale - Parent Version | through study completion, an average of 6 month
  Is a 12-item measure that assesses a child's prosocial behaviors, communication skills, and self control.Each item on this Scale states a behavior that a child may display in a social setting. The parent assesses how well each statement describes the child. Responses are coded on a five-point Likert scale ranging from zero (Not at all) to 4 (Very Well). The Scale contains two subscales: Prosocial/Communication Skills (Items 4, 7, 9, 10, 11 and 12) and Emotional Regulation Skills (Items 1, 2, 3, 5, 6, and 8). In addition to the subscale scores, a total score on the 12 items is also reported. T-tests of means for subscale scores and for the total score on this Scale show significant differences between the normative and control groups. The internal consistency measure (Cronbach alpha values) indicates that the total score and subscale scores are useful.
Behavioral problems and psychological assessment: The Strengths and Difficulties Questionnaire (SDQ). | through study completion, an average of 6 month
  This 25-question questionnaire explores different symptoms grouped into 5 sub-scales (with 5 items each): (1) emotional symptoms, (2) behavioral problems, (3) problems with peers, (4) symptoms of lack of attention and hyperactivity, and (5) prosocial skills. The first four sub-scales refer to difficulties that children may have and may be grouped together in a general sub-scale of difficulties (20 items). The sub-scale of prosocial skills refers to positive and adaptive behaviours in relationships with others. Each item is answered on a scale of responses from 1=not true to 3=absolutely true. There is a version for Educators, parents (to evaluate children from 4 to 16 years old), and a self-report for teenagers (ages 11 to 16 years old). It has been widely used and has shown good psychometric characteristics. The Educators' and parents' version of this instrument will be used. The higher score the better the skill.
Behavioral problems and psychological assessment: The Eyberg Child Behavior Inventory (ECBI) | through study completion, an average of 6 month
  The ECBI is a behaviorally specific rating scale that assesses the current frequency and severity of disruptive behaviors in the home setting, as well as the extent to which parents find the behavior troublesome. By evaluating the variety and frequency of behaviors commonly exhibited by all children, the instrument distinguishes normal behavior problems from conduct-disordered behavior in children and adolescents. This instrument requires the project pay a license per each time it is responded. The higher score the better the skill.
Empathy Scale for Children | through study completion, an average of 6 month
  Empathy Scale for Children (ESC) is a tool which is developed for measuring children's empathic skills. The scale consists of picture cards about four basic emotions (happiness, sadness, anger and fear) and cards about facial expressions. The higher score the better the skill.
The Tower of London | through study completion, an average of 6 month
  Its objective is to evaluate cognitive planning. The Tower of London was developed by Shallice (1982), based on the pre-existing Tower of Hanoi. This instrument is applied to children through individual interviews. The participants' task is to convert the initial position of the balls to the position demonstrated by the evaluator. Ball movements are limited by the fact that pegs differ in terms of the maximum number of balls they can hold at any time, and participants cannot move more than one ball at a time. The higher score the better the skill.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete, MD, PhD, Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data about primary and secondary outcomes without identifiable variables such as name, date of birth, or others.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study and until five years after the end of the study.
Access Criteria: Any researchers who ask the principal investigator fot secondary analysis, data anonymized.
URL: https://www.ismeuandes.cl/

REFERENCES:
- [Background] Sawyer SM, Azzopardi PS, Wickremarathne D, Patton GC. The age of adolescence. Lancet Child Adolesc Health. 2018 Mar;2(3):223-228. doi: 10.1016/S2352-4642(18)30022-1. Epub 2018 Jan 30. PMID 30169257
- [Background] Aldington S, Williams M, Nowitz M, Weatherall M, Pritchard A, McNaughton A, Robinson G, Beasley R. Effects of cannabis on pulmonary structure, function and symptoms. Thorax. 2007 Dec;62(12):1058-63. doi: 10.1136/thx.2006.077081. Epub 2007 Jul 31. PMID 17666437
- [Background] Weiser M, Zarka S, Werbeloff N, Kravitz E, Lubin G. Cognitive test scores in male adolescent cigarette smokers compared to non-smokers: a population-based study. Addiction. 2010 Feb;105(2):358-63. doi: 10.1111/j.1360-0443.2009.02740.x. Epub 2009 Nov 17. PMID 19919595
- [Background] Winward JL, Hanson KL, Bekman NM, Tapert SF, Brown SA. Adolescent heavy episodic drinking: neurocognitive functioning during early abstinence. J Int Neuropsychol Soc. 2014 Feb;20(2):218-29. doi: 10.1017/S1355617713001410. PMID 24512674
- [Background] Solowij N, Jones KA, Rozman ME, Davis SM, Ciarrochi J, Heaven PC, Lubman DI, Yucel M. Verbal learning and memory in adolescent cannabis users, alcohol users and non-users. Psychopharmacology (Berl). 2011 Jul;216(1):131-44. doi: 10.1007/s00213-011-2203-x. Epub 2011 Feb 17. PMID 21328041
- [Background] Servicio Nacional para la Prevención y Rehabilitación del Consumo de Drogas y Alcohol. Décimo Segundo Estudio Nacional de Drogas en Población Escolar de Chile 2017 [Available from: https://www.senda.gob.cl/wp-content/uploads/2019/01/ENPE-2017.pdf.
- [Background] Meier MH, Caspi A, Ambler A, Harrington H, Houts R, Keefe RS, McDonald K, Ward A, Poulton R, Moffitt TE. Persistent cannabis users show neuropsychological decline from childhood to midlife. Proc Natl Acad Sci U S A. 2012 Oct 2;109(40):E2657-64. doi: 10.1073/pnas.1206820109. Epub 2012 Aug 27. PMID 22927402
- [Background] Medina Cardenas E, Dobert Versin MT. [Chile: program for the primary prevention of alcoholism in schools]. Bol Oficina Sanit Panam. 1981 Feb;90(2):95-104. No abstract available. Spanish. PMID 6452149
- [Background] National Council for Narcotics Control. Catálogo de Publicaciones CONACE 2000-2009 2010 [Available from: https://bibliodrogas.gob.cl/biblioteca/documentos/DROGAS_CL_6192.PDF.
- [Background] National Service for the Prevention and Rehabilitation of Substance and Alcohol Use. Programa Continuo Preventivo 2021 [Available from: https://www.senda.gob.cl/prevencion/iniciativas/prevencion-escolar/programa-continuo-preventivo/.
- [Background] Corea V ML, Zubarew G T, Valenzuela M MT, Salas P F. [Evaluation of the program "Strong families: love and limits" in families with teenagers aged 10 to 14 years]. Rev Med Chil. 2012 Jun;140(6):726-31. doi: 10.4067/S0034-98872012000600005. Spanish. PMID 23282609
- [Background] National Council for Narcotics Control. Estrategia Nacional de Drogas y Alcohol 2011-2014 2011 [Available from: http://www.cicad.oas.org/fortalecimiento_institucional/planesnacionales/docs/estrategia_drogas_alcohol.pdf.
- [Background] R. J, Harris J, Skoog A. A review of classroom-based SEL programs at the middle school level. In: The Guilford Press, editor. Handbook of social and emotional learning: Research and practice2015. p. 167-80.
- [Background] Perry CL, Williams CL, Veblen-Mortenson S, Toomey TL, Komro KA, Anstine PS, McGovern PG, Finnegan JR, Forster JL, Wagenaar AC, Wolfson M. Project Northland: outcomes of a communitywide alcohol use prevention program during early adolescence. Am J Public Health. 1996 Jul;86(7):956-65. doi: 10.2105/ajph.86.7.956. PMID 8669519
- [Background] Komro KA, Perry CL, Veblen-Mortenson S, Farbakhsh K, Toomey TL, Stigler MH, Jones-Webb R, Kugler KC, Pasch KE, Williams CL. Outcomes from a randomized controlled trial of a multi-component alcohol use preventive intervention for urban youth: project northland Chicago. Addiction. 2008 Apr;103(4):606-18. doi: 10.1111/j.1360-0443.2007.02110.x. Epub 2008 Feb 4. PMID 18261193
- [Background] Gol-Guven M. The effectiveness of the Lions Quest Program: Skills for Growing on school climate, students' behaviors, perceptions of school, and conflict resolution skills. European Early Childhood Education Research Journal. 2017;25(4):575-94.
- [Background] Eisen M, Zellman GL, Murray DM. Evaluating the Lions-Quest "Skills for Adolescence" drug education program. Second-year behavior outcomes. Addict Behav. 2003 Jul;28(5):883-97. doi: 10.1016/s0306-4603(01)00292-1. PMID 12788263
- [Background] Catalano RF, Haggerty KP, Oesterle S, Fleming CB, Hawkins JD. The importance of bonding to school for healthy development: findings from the Social Development Research Group. J Sch Health. 2004 Sep;74(7):252-61. doi: 10.1111/j.1746-1561.2004.tb08281.x. No abstract available. PMID 15493702
- [Background] Hawkins JD, Catalano RF, Kosterman R, Abbott R, Hill KG. Preventing adolescent health-risk behaviors by strengthening protection during childhood. Arch Pediatr Adolesc Med. 1999 Mar;153(3):226-34. doi: 10.1001/archpedi.153.3.226. PMID 10086398
- [Background] Brown EC, Catalano RF, Fleming CB, Haggerty KP, Abbott RD. Adolescent substance use outcomes in the Raising Healthy Children project: a two-part latent growth curve analysis. J Consult Clin Psychol. 2005 Aug;73(4):699-710. doi: 10.1037/0022-006X.73.4.699. PMID 16173857
- [Background] Catalano RF, Mazza JJ, Harachi TW, Abbott RD, Haggerty KP, Fleming CB. Raising healthy children through enhancing social development in elementary school: Results after 1.5 years. Journal of School Psychology. 2003;41(2):143-64.
- [Background] Faggiano F, Galanti MR, Bohrn K, Burkhart G, Vigna-Taglianti F, Cuomo L, Fabiani L, Panella M, Perez T, Siliquini R, van der Kreeft P, Vassara M, Wiborg G; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: EU-Dap cluster randomised controlled trial. Prev Med. 2008 Nov;47(5):537-43. doi: 10.1016/j.ypmed.2008.06.018. Epub 2008 Jul 9. PMID 18657569
- [Background] Faggiano F, Vigna-Taglianti F, Burkhart G, Bohrn K, Cuomo L, Gregori D, Panella M, Scatigna M, Siliquini R, Varona L, van der Kreeft P, Vassara M, Wiborg G, Galanti MR; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: 18-month follow-up of the EU-Dap cluster randomized controlled trial. Drug Alcohol Depend. 2010 Apr 1;108(1-2):56-64. doi: 10.1016/j.drugalcdep.2009.11.018. Epub 2010 Jan 18. PMID 20080363
- [Background] Bond L, Patton G, Glover S, Carlin JB, Butler H, Thomas L, Bowes G. The Gatehouse Project: can a multilevel school intervention affect emotional wellbeing and health risk behaviours? J Epidemiol Community Health. 2004 Dec;58(12):997-1003. doi: 10.1136/jech.2003.009449. PMID 15547059
- [Background] McNeely C, Falci C. School connectedness and the transition into and out of health-risk behavior among adolescents: a comparison of social belonging and teacher support. J Sch Health. 2004 Sep;74(7):284-92. doi: 10.1111/j.1746-1561.2004.tb08285.x. No abstract available. PMID 15493705
- [Background] Irvin MJ, Meece JL, Byun SY, Farmer TW, Hutchins BC. Relationship of school context to rural youth's educational achievement and aspirations. J Youth Adolesc. 2011 Sep;40(9):1225-42. doi: 10.1007/s10964-011-9628-8. Epub 2011 Jan 28. PMID 21755376
- [Background] Gaete J, Olivares E, Rojas-Barahona CA, Labbe N, Rengifo M, Silva M, Lepe L, Yanez C, Chen MY. [Factors associated with health promoting behaviors among Chilean adolescents]. Rev Med Chil. 2014 Apr;142(4):418-27. doi: 10.4067/S0034-98872014000400002. Spanish. PMID 25117031
- [Background] Shochet IM, Smith CL, Furlong MJ, Homel R. A prospective study investigating the impact of school belonging factors on negative affect in adolescents. J Clin Child Adolesc Psychol. 2011;40(4):586-95. doi: 10.1080/15374416.2011.581616. PMID 21722030
- [Background] Stallard P, Spears M, Montgomery AA, Phillips R, Sayal K. Self-harm in young adolescents (12-16 years): onset and short-term continuation in a community sample. BMC Psychiatry. 2013 Dec 2;13:328. doi: 10.1186/1471-244X-13-328. PMID 24294921
- [Background] Ream RK, Rumberger RW. Student engagement, peer social capital, and school dropout among Mexican American and non-Latino white students. Sociology of education. 2008;81(2):109-39.
- [Background] Demanet J, Van Houtte M. School belonging and school misconduct: the differing role of teacher and peer attachment. J Youth Adolesc. 2012 Apr;41(4):499-514. doi: 10.1007/s10964-011-9674-2. Epub 2011 May 13. PMID 21567214
- [Background] West* P, Sweeting H, Leyland A. School effects on pupils' health behaviours: evidence in support of the health promoting school. Research papers in Education. 2004;19(3):261-91.
- [Background] Weissberg R, Caplan M, Bennetto L, Jackson A. The New Haven Social Development Program: Sixth-grade social problem-solving model. New Haven, CT: Yale University. 1990.
- [Background] Caplan M, Weissberg R. The New Haven Social Development Program: Sixth-grade substance use prevention module. Chicago: University of Illinois at Chicago. 1990.
- [Background] Caplan M, Weissberg RP, Grober JS, Sivo PJ, Grady K, Jacoby C. Social competence promotion with inner-city and suburban young adolescents: effects on social adjustment and alcohol use. J Consult Clin Psychol. 1992 Feb;60(1):56-63. doi: 10.1037//0022-006x.60.1.56. PMID 1556286
- [Background] Weissberg RP, Barton HA, Shriver TP. The Social-Competence Promotion Program for Young Adolescents. 1997.
- [Background] The Oregon Addiction and Mental Health Services. Social Competence Promotion Program for Young Adolescents (SCPP-YA) 2012 [Available from: https://www.theathenaforum.org/social_competence_promotion_program_for_young_adolescents_scpp_ya.
- [Background] Brigham GS, Feaster DJ, Wakim PG, Dempsey CL. Choosing a control group in effectiveness trials of behavioral drug abuse treatments. J Subst Abuse Treat. 2009 Dec;37(4):388-97. doi: 10.1016/j.jsat.2009.05.004. Epub 2009 Jun 23. PMID 19553062
- [Background] Junta Nacional de Auxilio Escolar y BecasDirección Nacional. SINAESistema Nacional de Asignación conEquidad para Becas JUNAEB 2005 [Available from: https://www.junaeb.cl/wp-content/uploads/2013/02/libro_junaeb.pdf.
- [Background] Ramirez S, Gana S, Godoy MI, Valenzuela D, Araya R, Gaete J. Validation of the European Drug Addiction Prevention Trial Questionnaire (EU-Dap) for substance use screening and to assess risk and protective factors among early adolescents in Chile. PLoS One. 2021 Oct 11;16(10):e0258288. doi: 10.1371/journal.pone.0258288. eCollection 2021. PMID 34634082
- [Background] Sorsdahl K, Stein DJ, Myers B. Psychometric properties of the Social Problem Solving Inventory-Revised Short-Form in a South African population. Int J Psychol. 2017 Apr;52(2):154-162. doi: 10.1002/ijop.12192. Epub 2015 Aug 7. PMID 26249118
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559
- [Background] Pastor MC, Lopez-Penades R, Cifre E, Moliner-Urdiales D. The Spanish Version of the Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): A Psychometric Evaluation in Early Adolescence. Span J Psychol. 2019 May 31;22:E30. doi: 10.1017/sjp.2019.30. PMID 31148532
- [Background] Gaete J, Montero-Marin J, Valenzuela D, Rojas-Barahona CA, Olivares E, Araya R. Mental health among children and adolescents: Construct validity, reliability, and parent-adolescent agreement on the 'Strengths and Difficulties Questionnaire' in Chile. PLoS One. 2018 Feb 5;13(2):e0191809. doi: 10.1371/journal.pone.0191809. eCollection 2018. PMID 29401472
- [Background] Gaete J, Montero-Marin J, Rojas-Barahona CA, Olivares E, Araya R. Validation of the Spanish Version of the Psychological Sense of School Membership (PSSM) Scale in Chilean Adolescents and Its Association with School-Related Outcomes and Substance Use. Front Psychol. 2016 Dec 6;7:1901. doi: 10.3389/fpsyg.2016.01901. eCollection 2016. PMID 27999554
- [Background] U.S. Food & Drug Administration. Regulations: Good Clinical Practice and Clinical Trials [Available from: https://www.fda.gov/science-research/clinical-trials-and-human-subject-protection/regulations-good-clinical-practice-and-clinical-trials.
- [Background] Guzman J, Kessler RC, Squicciarini AM, George M, Baer L, Canenguez KM, Abel MR, McCarthy A, Jellinek MS, Murphy JM. Evidence for the effectiveness of a national school-based mental health program in Chile. J Am Acad Child Adolesc Psychiatry. 2015 Oct;54(10):799-807.e1. doi: 10.1016/j.jaac.2015.07.005. Epub 2015 Aug 3. PMID 26407489
- [Background] Gaete J, Valenzuela D, Rojas-Barahona C, Valenzuela E, Araya R, Salmivalli C. The KiVa antibullying program in primary schools in Chile, with and without the digital game component: study protocol for a randomized controlled trial. Trials. 2017 Feb 20;18(1):75. doi: 10.1186/s13063-017-1810-1. PMID 28219403
- [Background] Thorisdottir IE, Asgeirsdottir BB, Kristjansson AL, Valdimarsdottir HB, Jonsdottir Tolgyes EM, Sigfusson J, Allegrante JP, Sigfusdottir ID, Halldorsdottir T. Depressive symptoms, mental wellbeing, and substance use among adolescents before and during the COVID-19 pandemic in Iceland: a longitudinal, population-based study. Lancet Psychiatry. 2021 Aug;8(8):663-672. doi: 10.1016/S2215-0366(21)00156-5. Epub 2021 Jun 3. PMID 34090582
- [Background] Social competence - parent - fast track project. (2022, May 1). Fast Track Project. https://fasttrackproject.org/measure/social-competence-parent/
- [Derived] Gaete J, Ramirez S, Rojas-Barahona CA, Romo V, Rios N, Araya R. Japi 2.0, a gaming platform to stimulate cognitive and non-cognitive skills in early childhood: protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2025 Jan 11;11(1):5. doi: 10.1186/s40814-025-01593-w. PMID 39799357